CLINICAL TRIAL: NCT00900679
Title: A Standardized Nursing Intervention Protocol for Ovarian Cancer as a Chronic Illness
Brief Title: Effects of a Teaching Intervention With an Advanced Practice Nurse on Quality of Life and Psychosocial and Symptom Distress in Patients With Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Marcia Grant, City of Hope Comprehensive Cancer Center
Other Study IDs: 08032; P30CA033572 (NIH); CHNMC-08032; CDR0000629411 (Registry Identifier: PDQ)
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Ovarian Cancer; Transitional Care Planning
Keywords: transitional care planning; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Counseling; Early Intervention, Educational; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: telephone-based intervention
Other: counseling intervention
Other: educational intervention
Other: medical chart review
Other: questionnaire administration
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: A teaching intervention with an advanced practice nurse may help reduce psychosocial and symptom distress and improve the well-being and quality of life of patients with ovarian cancer.

PURPOSE: This clinical trial is studying the effects of a teaching intervention with an advanced practice nurse on quality of life and psychosocial and symptom distress in patients with ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the effects of a standardized nursing intervention protocol (SNIP) model with an advanced practice nurse vs usual care on overall quality of life and psychological distress from initial treatment to 6 months after diagnosis in patients with ovarian cancer.
* To compare symptom control in these patients.
* To compare geriatric assessment outcomes in these patients.
* To compare the effects of the SNIP intervention vs usual care on resource use by these patients.
* To test the effects of SNIP on patients' and clinicians' satisfaction with care.
* To describe the effects of SNIP on management of transitions from one phase of chronic illness to another.
* To identify subgroups of patients with ovarian cancer who benefit most from the SNIP in relation to sociodemographic characteristics, disease/treatment factors, and geriatric assessment predictors.
* To obtain feedback from clinicians regarding interpretation of findings and application to the routine care of ovarian cancer patients.

OUTLINE: Patients are stratified according to age (18 to 60 years vs 61 years and over). Patients are sequentially enrolled into 1 of 2 groups. Patients are initially enrolled in group I. Once enrollment in group I is completed, additional patients are enrolled in group II.

* Group I (usual care): Patients complete questionnaires, including the FACT-Ovarian, Memorial Symptom Assessment Scale, Psychological Distress Thermometer, and Comprehensive Geriatric Assessment, at baseline and at 3 and 6 months. Clinicians also complete questionnaires, including the Clinician Satisfaction with Intervention Questionnaire. Patients' medical charts are reviewed to collect information about treatment, episodes of care, and readmissions.
* Group II (advanced practice nurse [APN] intervention): Patients undergo face-to-face individualized teaching sessions with an APN twice a month for 2 months. The sessions focus on the patient's physical, psychological, social, and spiritual well-being and the content is tailored to the patient's preferences and needs. Patients are then contacted by the APN via telephone once a month for 4 months to clarify questions and content from the teaching sessions, review any patient concerns, including concerns associated with a transition, and coordinate interdisciplinary resources, including community resources, as needed. Patients and clinicians complete questionnaires as in group I. Patients' medical charts are also reviewed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ovarian cancer (any stage)

PATIENT CHARACTERISTICS:

* Lives within a 30-mile radius of City of Hope National Medical Center
* No prior cancer

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Quality of life, psychological distress, symptom control, geriatric assessment outcome, and resource use at 3 months
Quality of life, psychological distress, symptom control, geriatric assessment outcome, and resource use at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Grant, RN, DNSc, FAAN, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States